CLINICAL TRIAL: NCT05753020
Title: A Pilot Study of The CKM JumpStart Tool
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Susan Wong, Associate Professor: School of Medicine, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: STUDY00017195
Record Dates: First submitted 2023-02-21; First posted 2023-03-03 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Chronic Kidney Diseases
Keywords: Kidney supportive care; Communication; Shared decision-making; Conservative kidney management; Palliative care; End-of-life care
MeSH Terms: conditions — Renal Insufficiency, Chronic; Communication

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CKM Jumpstart Tool (Experimental): Receives intervention
  Interventions: Behavioral: CKM Jumpstart Tool
- Control (No Intervention): Does not receive intervention

INTERVENTIONS:
Behavioral: CKM Jumpstart Tool — The CKM JumpStart Tool is a 1-page handout that describes the values of a patient and words that a providers can try with the patient to explore the patient' values more and to provide a values-based introduction to CKM. The values described in the CKM JumpStart Tool is based on a patient's response to a single validated question that we will ask the patient at T1, if they had to choose, do they value care directed at longevity or comfort. Using the patient's answer to the values question, study staff will generate a CKM JumpStart Tool prior to their upcoming clinic visit with their nephrologist. Study staff will inform the patient that their response to the values question will be shared with their provider prior to their next clinic visit and that their providers might bring up their values and treatment options for kidney disease, if the situation permits. We will share the CKM Jumpstart Tool with their provider and provide instruction on how to use the Tool.
  Arms: CKM Jumpstart Tool

SUMMARY:
This is a randomized pilot study to test the feasibility and acceptability of a tool to promote discussion about conservative kidney management (CKM) among older patients with advanced CKD and their providers.

DETAILED DESCRIPTION:
This study is a randomized pilot study to test the acceptability and feasibility of a novel communication tool, called the CKM Jumpstart Tool, to promote discussion of CKM between patients with advanced CKM and their healthcare providers, the investigators hypothesize that the Guide will be feasible and acceptable to patients and their healthcare providers as reflected in greater discussion of CKM between them following use of the Tool as compared with usual care. The investigators will enroll 76 patients aged 75 years and older with advanced CKD and their healthcare providers from University of Washington Medicine and Veterans Affairs Puget Sound Health Care System. Patients will be randomized together in a 1:1 fashion to receive the intervention or usual care. Data from participants will be collected at the time of enrollment (T1), within 2-weeks of their following clinic visit with their healthcare provider (T2), and approximately 3-month after this clinic visit (T3). The primary outcome measure and measure of feasibility is difference in patient-reported rates of discussion of CKM with a healthcare provider at T2 and T3. The investigators will also evaluate whether provider document in the medical chart of patients whether they had a discussion about CKM with the patient at T2 and T3. The investigators will also collect attrition rates at T2 and T3 as a measure of acceptability. The investigators will further assess user experience of the CKM JumpStart by performing a qualitative analysis of post-intervention interviews with patients and nephrologists, coding for themes elucidating pros, cons and other considerations with using the CKM JumpStart Tool and discussion about CKM.

ELIGIBILITY:
Patients

Inclusion:

* Adults aged ≥75 years
* Advanced CKD as defined as having at least 2 outpatient measures of eGFR <25 ml/min/1.73m2 separated by >90 days in the prior year and with at least 1 eGFR measure <20.
* English-speaking
* Receive care from a provider at UW Medicine or VA Puget Sound
* Open to discussing their values and treatment options for kidney disease with their provider.

Exclusion:

* Unable to complete the informed consent process
* Currently receiving maintenance dialysis

Providers Inclusion

* Their patient is a participant in the study.
* Are a UW Medicine or VA Puget Sound provider or trainee.

Exclusion

• None

Min Age: 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Gender Based: Yes — self-representation
Enrollment: 76 (Estimated)
Dates: Start 2023-04-10 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Patient-provider discussion of CKM | 3 months
  We will ask patients whether they had discussed CKM with their healthcare provider at T2 and T3.
Attrition | 3 months
  We will record the proportion of participants in each study arm who withdraw from the study and the reasons why at T2 and T3. Study withdrawal would indicate that the Tool and/or study is unacceptable or burdensome to the participant.

SECONDARY OUTCOMES:
Treatment preference | 3 months
  At each study visit, we will record each patient's preference for dialysis or CKM using the Decision Conflict Scale at each study visit.
Quality of Communication | 3 months
  At each study visit, patients will be asked to rate the quality of serious illness communication with their nephrologists using the Quality of Communication Questionnaire.
Documentation of CKM Discussion | 3 months
  At T2 and T3, we will review each patient's recent nephrology clinic notes to determine whether their providers documented a discussion with patients about CKM.
Patient Post-Intervention Interview | 2 weeks
  For patients randomized to receive the intervention, at T2, patients will be invited to answer 4 open-ended questions about their clinical encounter with their provider. Questions will pertain to topics discussed during the encounter with their provider, whether their provider asked them about their values, whether CKM was discussed, and their perception of CKM based on the conversation.
Provider Use of CKM Jumpstart Tool | 2 weeks
  For patients randomized to receive the intervention, at T2, their providers will be asked whether they had used the CKM Jumpstart Tool during their visit, and if not their reasons for not using the Tool.

CONTACTS AND LOCATIONS:
Overall Officials: Susan P Wong, MD, MS, Principal Investigator — University of Washington
Locations (2):
- United States (2):
  - VA Puget Sound Health Care System, Seattle, Washington
  - University of Washington, Seattle, Washington

DOCUMENTS (1):
  • Study Protocol (2023-02-15): https://cdn.clinicaltrials.gov/large-docs/20/NCT05753020/Prot_000.pdf